CLINICAL TRIAL: NCT00124241
Title: A Phase IIb Extension Study of LdT (Telbivudine), Lamivudine or LdT Plus Lamivudine in Patients With Chronic Hepatitis B Who Have Completed Study NV-02B-003
Brief Title: An Extension Study of Telbivudine, Lamivudine or Telbivudine Plus Lamivudine in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV-02B-010
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Telbivudine; Lamivudine

INTERVENTIONS:
Drug: telbivudine
Drug: lamivudine

SUMMARY:
This is an extension study for patients who have previously completed Idenix Study NV-02B-003. This study is being conducted to compare the safety and effectiveness of treatment beyond 1 year of telbivudine and telbivudine combined with lamivudine, a drug currently approved for the treatment of hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed protocol NV-02B-003 without a serious adverse event attributed to study drug
* Patient remains seropositive for hepatitis B surface antigen (HBsAg)

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breast-feeding
* Patient has signs of decompensated chronic hepatitis B

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2003-02 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Los Angeles, California, United States
- Toronto, Canada
- Hong Kong, China
- Paris, France